CLINICAL TRIAL: NCT03879343
Title: The Prevalence and Predictors of Gastrointestinal Symptoms in Children With Attention Deficit / Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG SIU FUNG JONATHAN, Principal investigator, Hospital Authority, Hong Kong
Other Study IDs: 2018.285
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Gastrointestinal Diseases
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical group: Children aged six to eleven with clinical diagnosis of attention deficit / hyperactivity disorder were recruited for interview and completion of questionnaires
  Interventions: Other: Known diagnosis of attention deficit / hyperactivity disorder
- Control group: Normally developing children aged six to eleven studying in local mainstream primary schools were recruited for completion of questionnaires

INTERVENTIONS:
Other: Known diagnosis of attention deficit / hyperactivity disorder — Clinical group includes subjects with clinical diagnosis of attention deficit / hyperactivity disorder
  Groups: Clinical group

SUMMARY:
This study is to examine the gut problems in children with attention deficit hyperactivity disorders (ADHD) and is conducted by the Department of Psychiatry of Alice Ho Miu Ling Nethersole Hospital. Children with ADHD who attend our department will be recruited with their parents/guardians' consent. Only the primary caregiver will be invited for an interview to assess the recruited children's gut problems, autistic features, emotional problems, diet pattern and medical history. The data will be compared with normal children who are recruited as control in local primary schools. The aim of this study is to know whether children with ADHD have higher chance of gut problems, and to assess other factors associated with the linkage.

ELIGIBILITY:
Inclusion Criteria:

* The study group will be recruited if the following criteria are met:

  1. Aged 6 to 11 years old
  2. Children with a diagnosis of ADHD made by psychiatrists according to Diagnostic and Statistical Manual for Mental Disorder, fifth edition criteria
  3. Currently study in mainstream schools in Hong Kong

The control group will be recruited if the following criteria are met:

1. Age 6 to 11 years old
2. Currently study in mainstream schools in Hong Kong
3. Typically developing in good mental and physical health

Exclusion Criteria:

* For both groups, the participant will be excluded if the following criterion is met:

  1. Children who are suffering from mental retardation
  2. Children who are suffering from organic illnesses that affect gastrointestinal function
  3. Children who are suffering from severe mental illnesses
  4. Children who have ever received, or are currently on, medication for ADHD
  5. Children who are currently taking medication for illnesses other than ADHD
  6. Primary caregiver does not understand Chinese

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will recruit children who attend a local district child and adolescent psychiatry outpatient department during the study period. A consecutively selected sample of participants is recruited until it reaches the target number of sample size. The normal controls will be recruited via primary schools.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The number of children with ADHD had gastrointestinal (GI) symptoms | One month prior to interview
  Functional gastrointestinal symptoms as measured by Rome IV Diagnostic Questionnaire on Pediatric Functional Gastrointestinal Disorders (R4PGD)

SECONDARY OUTCOMES:
The number of children with ADHD had GI symptoms after controlling for the potential confounding factors including co-morbid autism spectrum disorder (ASD) symptoms, emotional symptoms and diet pattern | One month prior to interview

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Siu Fung Ng, Principal Investigator — Hospital Authority, Hong Kong
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Tai Po, New Territories, Hong Kong